CLINICAL TRIAL: NCT07050628
Title: Long-Term Tracking of Fluid Dynamics in Cerebrospinal Fluid Shunts With a Wireless Thermal Anisotropy Measurement Device During Activities of Daily Living Including Sleep
Brief Title: Assessment of CSF Shunt Flow During Activities of Daily Living and Sleep With a Thermal Measurement Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhaeos, Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-03; 5UG3NS130338 (NIH)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- No Recent Revision (Experimental): Pediatric hydrocephalus patients with an existing ventricular CSF shunt and a history of stable ventricular size, no shunt revision in the previous 2 years, and no current symptoms of shunt failure will be enrolled.
  Interventions: Device: wireless thermal anisotropy measurement device
- Recent Revision (Experimental): Pediatric hydrocephalus patients with an existing ventricular CSF shunt and a shunt revision in the previous 7 days who the investigator judges will likely be discharged within 4 days of the enrollment date will be enrolled.
  Interventions: Device: wireless thermal anisotropy measurement device

INTERVENTIONS:
Device: wireless thermal anisotropy measurement device — Wireless wearable thermal anisotropy measurement device designed for use at home

SUMMARY:
This study evaluates the performance of a device for non-invasively assessing cerebrospinal fluid (CSF) shunt flow over multiple measurements performed by a study subject during activities of daily living and sleep

ELIGIBILITY:
Inclusion Criteria:

1. Existing ventricular CSF shunt
2. (Cohort A) A history of stable ventricular size, no shunt revision in the previous 2 years, and no current symptoms of shunt failure
3. (Cohort B) A shunt revision in the previous 7 days and the investigator judges that the patient will likely be discharged within 4 days of the enrollment date
4. Region of intact skin overlying an unambiguously identifiable palpable chronically indwelling ventricular shunt which crosses the clavicle and is appropriate in size for application of the study device
5. Signed informed consent by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
6. Subject is at least 5 years old but < 22 years old

Exclusion Criteria:

1. Shunt is not palpable or depth of shunt where the device will be placed is greater than 4 mm per ultrasound evaluation
2. Presence of an interfering open wound or edema in the study device measurement region
3. Subject-reported history of serious adverse skin reactions to silicone-based adhesives
4. Investigator judges that the subject is likely to be lost to follow-up due to unavailability or clinical outcome being unobtainable
5. Investigator judges that the subject is unlikely to successfully take reliable measurements at home
6. Investigator judges that the subject/subject's caretaker would not be able to successfully place the device without assistance
7. Use of the study device would interfere with standard patient care, or emergency surgery that cannot be delayed, or participation in the study will interfere with, or be detrimental to, administration of optimal healthcare to the subject
8. Prior enrollment in this study
9. Participation in any other investigational procedural, pharmaceutical, and/or device study that may influence the collection of valid data under this study

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Device Effects | 30 days
  The co-primary endpoints in this study are the rate of ADEs and SADEs that occur per wear hour.

SECONDARY OUTCOMES:
ADEs and SADEs per wear period | 30 days
  rate of ADEs and SADEs per wear period
ADEs and SADEs per subject | 30 days
  rate of ADEs and SADEs per subject;
ADEs and SADEs that preclude the continued use of the study device | 30 days
  rate of ADEs and SADEs that preclude the continued use of the study device
Device deficiencies resulting in incomplete monitoring data | 30 days
  percent of device deficiencies resulting in incomplete monitoring data
Local skin reactions per wear session; | 30 days
  number of local skin reactions per wear session;
Usability score | 30 days
  usability score based on post-study survey

CONTACTS AND LOCATIONS:
Locations (1):
- Rhaeos Inc., Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No